CLINICAL TRIAL: NCT03405012
Title: Understanding Changes in Treatment-related Regional Bone Turnover Using 18F-fluoride-PET/CT in HIV-1-infected Men: PETRAM Study
Brief Title: Regional Bone Turnover Using 18F-fluoride-PET/CT in HIV-1-infected Men: PETRAM Study
Acronym: PETRAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 16/0657
Record Dates: First submitted 2017-04-25; First posted 2018-01-19 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a 48 week study to explore the pathogenesis of HIV treatment related bone disease by using a novel imaging technique, 18F-Fluoride Positron Emission Tomography (18F-PET/CT), which measures regional bone formation. The study will include other standard methods (serum bone markers and DXA) for comparison. Patients enrolled will have baseline, week 24 and week 48 assessment, with baseline being the date of replacing tenofovir disoproxil fumarate (TDF) in their HIV treatment regimen with tenofavir alafenamide fumarate (TAF), compared to a control group continuing TDF. Allocation to change to TAF or continue TDF will be randomised to allow an unbiased assessment of bone changes.

DETAILED DESCRIPTION:
Study Design:

This is an observational, open-label, non-randomised, single centre, 48-week study to explore the utility of a novel scanning platform exploring bone turnover during an immediate or deferred (for 48 weeks) switch from Eviplera® to Odefsey® in HIV-1 infected men aged 40 years or older, and stable on Eviplera®.

Participants:

HIV-1-infected males, aged ≥40 years, on Eviplera® >24 weeks, with plasma HIV RNA (pVL) <50cp/mL and without any known history of osteoporosis.

Groups to be Compared: 1. HIV-1-infected males aged ≥40, stable on Eviplera® (rilpivirine (RPV)/emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF)) and remaining on EvipleraÒ for 48 weeks on study; 2. HIV-1-infected males aged ≥40 years, switched to Odefsey® (RPV/FTC/tenofovir alafenamide (TAF)) at study enrollment.

Study Hypothesis: We hypothesis that there will be ongoing subclinical loss of bone at the hip and lumbar spine as measured by 18F-fluoride-PET/CT in those remaining of Eviplera®, and in those switching to Odefsey® there will be reversal of some of this subclinical loss at 24 and 48 weeks post switch.

Primary Outcome Measure(s):To determine the change in regional bone formation at the hip and lumbar spine as measured by 18F-fluoride-PET/CT at 24 weeks post switch from Eviplera® to Odefsey®.

Secondary Outcome Measure(s): 1. Change in regional bone formation at the hip and lumbar spine as measured by 18F-fluoride-PET/CT at 48 weeks post switch from Eviplera® to Odefsey®; 2. Assess safety and tolerability of switching to Odefsey®; 3. To compare DXA changes at the hip and lumbar spine to those detected on 18F-fluoride-PET/CT; 4. Measure changes in plasma/serum bone biomarkers over 24 and 48 weeks; 5. To measure the changes in FRAX® score at week 48.

ELIGIBILITY:
INCLUSION CRITERIA

* HIV-1-infected men aged ≥40 years;
* Virologically suppressed (<50 cp/mL) on Eviplera® for >24 weeks;
* No known history of osteoporosis (defined as a T-score > -2.5 at the lumbar spine, femoral neck or total hip using DXA);
* Willing to switch immediately to OdefseyÒ or remain on EvipleraÒ for the duration of the study;
* No immediate toxicity reason in the opinion of the investigator to switch away from Eviplera;
* Willing to comply with study procedures.

EXCLUSION CRITERIA

* Contraindication to the receipt of TAF;
* Contraindication to 18F-fluoride-PET/CT scanning;
* Anticipated to require additional radiological imaging during the 48 weeks of study participation with a total cumulative radiation dose of >50 millisieverts (mSv);
* Current or previous treatment (within the prior 12 months) which can affect bone metabolism including systemic corticosteroids for >4 weeks and bisphosphonates;
* Hepatitis C coinfected.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The rationale for restricting this study to males is to avoid heterogeneity.
Study Population: HIV-1-infected men aged ≥40 years on ART regimen containing rilpivirine/tenofovir disoproxil fumarate/ emtricitabine for at least 6 months.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in regional bone formation at the hip and lumbar spine as measured by 18F-PET/CT at 24 weeks. | 24 weeks
  Regions of interest will be applied to various regions within the hip including but are not limited to the femoral neck, intertrochanteric region, trochanter and total proximal femur. Further regions of interest will be applied to each vertebral body, skull, pelvis and femoral shaft using the static scan for the calculation of standardised uptake values (SUV). At week 24

SECONDARY OUTCOMES:
The change in regional bone formation at the hip and lumbar spine as measured by 18F-PET/CT at 48 weeks in patients starting a TAF-based ART regimen | 48 weeks
  Regions of interest will be applied to various regions within the hip including but are not limited to the femoral neck, intertrochanteric region, trochanter and total proximal femur. Further regions of interest will be applied to each vertebral body, skull, pelvis and femoral shaft using the static scan for the calculation of standardised uptake values (SUV).
  measured by 18F-PET/CT at 48 weeks
Bone mineral density at the hip and lumbar spine measured by DXA vs. 18F-PET/CT; | 24 and 48 weeks
  Regions of interest will be applied to including but not limited to the femoral neck, intertrochanteric region, total hip, each lumbar vertebral body, and upper femoral shaft for the calculation of Ki which reflects regional bone perfusion and bone turnover and will be compared to results obtained Dual-energy x-ray absorptiometry (DXA) scans will be performed at baseline (Visit 1b), weeks 24 (Visit 2b) and 48 (Visit 3b) to evaluate the change in areal bone mineral density (BMD) (in g/cm2) in response to treatment at the lumbar spine (L1-L4), total hip, femoral neck and whole body using standard protocols.
The changes in bone biomarkers over 24 and 48 weeks with changes in 18F-PET/CT; | 24 and 48 weeks
  Regions of interest will be applied to including but not limited to the femoral neck, intertrochanteric region, total hip, each lumbar vertebral body, and upper femoral shaft for the calculation of Ki which reflects regional bone perfusion and bone turnover, with changes in bone biomarkers. The bone markers to be analysed include, but are not limited to, procollagen Type I N terminal propeptide (PINP), and cross-linked C telopeptides of Type I collagen (CTX).

CONTACTS AND LOCATIONS:
Locations (1):
- Mortimer Market Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frost ML, Cook GJ, Blake GM, Marsden PK, Benatar NA, Fogelman I. A prospective study of risedronate on regional bone metabolism and blood flow at the lumbar spine measured by 18F-fluoride positron emission tomography. J Bone Miner Res. 2003 Dec;18(12):2215-22. doi: 10.1359/jbmr.2003.18.12.2215. PMID 14672357
- [Result] Cassetti I, Madruga JV, Suleiman JM, Etzel A, Zhong L, Cheng AK, Enejosa J; Study 903E Team*. The safety and efficacy of tenofovir DF in combination with lamivudine and efavirenz through 6 years in antiretroviral-naive HIV-1-infected patients. HIV Clin Trials. 2007 May-Jun;8(3):164-72. doi: 10.1310/hct0803-164. PMID 17621463
- [Result] Cook GJ, Lodge MA, Blake GM, Marsden PK, Fogelman I. Differences in skeletal kinetics between vertebral and humeral bone measured by 18F-fluoride positron emission tomography in postmenopausal women. J Bone Miner Res. 2000 Apr;15(4):763-9. doi: 10.1359/jbmr.2000.15.4.763. PMID 10780868
- [Result] Frost ML, Cook GJ, Blake GM, Marsden PK, Fogelman I. The relationship between regional bone turnover measured using 18F-fluoride positron emission tomography and changes in BMD is equivalent to that seen for biochemical markers of bone turnover. J Clin Densitom. 2007 Jan-Mar;10(1):46-54. doi: 10.1016/j.jocd.2006.10.006. Epub 2006 Dec 27. PMID 17289526